CLINICAL TRIAL: NCT00358683
Title: Open Label Long Term Clinical Trial Evaluating Safety of Chronic Therapy With Certolizumab Pegol, a PEGylated Fab Fragment of Humanized Antibody to Tumor Necrosis Factor Alpha (TNF) in Patients Suffering From Crohn's Disease and Having Completed C87055 Study.
Brief Title: A Trial Evaluating Safety of Chronic Therapy With Certolizumab Pegol in Crohn's Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C87069; RPCE06G0406
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Crohn's Disease
Keywords: certolizunab pegol; long term safety follow-up; Chrohn's disease; infliximab failures patients; Greek population
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

INTERVENTIONS:
Drug: Certolizumab pegol

SUMMARY:
The primary aim of this study is allow the patients suffering from Crohn's disease , who both completed the therapeutic confirmatory study C87055 of certolizumab pegol and benefited from the treatment, to receive treatment with certolizumab pegol until the drug is available for the Crohn's disease indication in Greece.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease diagnosis
* Patients having completed the treatment period of study C87055 (previously treated with infliximab) and benefited from the study treatment, as per investigatior's discretion.

Exclusion Criteria:

* Subject withdrawn prematurely from C87055 study.
* Subject who received treatment other than certolizumab pegol and other than medications permitted in C87055 study.
* Female patients of childbearing age who are NOT practicing (in the Investigator's opinion) effective birth control. All female patients must test negative on a serum pregnancy test before study entry and negative on urine testing immediately before every certolizumab pegol administration.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11

PRIMARY OUTCOMES:
For ethical reasons, provide the opportunity for patients > 18 years suffering from Crohn's disease who both completed the therapeutic confirmatory study C87055 of certolizumab pegol and benefited from the treatment, to receive treatment with certolizum

SECONDARY OUTCOMES:
Incidence of adverse events reported by the patients during the long-term treatment period of the study.

CONTACTS AND LOCATIONS:
Overall Officials: George Syrmalis, M.D. M.Sc. Ph.D., Study Director — UCB Pharma